CLINICAL TRIAL: NCT02230735
Title: Effectiveness of Bupivacaine With Epinephrine Injections Into the Uterosacral Ligaments for Post-operative Pain Control and the Use of Narcotic Pain Medication Following Robotic Assisted Total Hysterectomies
Brief Title: Bupivacaine Injections Into Uterosacral Ligaments During Robotic Assisted Total Hysterectomies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started.
Sponsor: Souza, Amanda, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SouzaA
Record Dates: First submitted 2014-08-12; First posted 2014-09-03 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Pain
Keywords: Robotic; Hysterectomy; Uterosacral; Bupivacaine; Robotic hysterectomy pain control
MeSH Terms: conditions — Pain | interventions — Epinephrine; Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipivacaine 0.5% with epinephrine (Experimental): Total of 14 ml of bupivacaine hydrochloride 0.5% with epinephrine 1:200,000, 7ml in right uterosacral ligament, 7ml in left uterosacral ligament
  Interventions: Drug: Bipivacaine 0.5% with epinephrine
- Normal Saline (Placebo Comparator): Total of 14 ml of normal saline, 7ml into the right uterosacral ligament and 7ml into the left uterosacral ligament
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bipivacaine 0.5% with epinephrine — Total of 14 ml of bupivacaine hydrochloride 0.5% with epinephrine 1:200,000, 7ml in right uterosacral ligament, 7ml in left uterosacral ligament
  Other Names: Marcaine With Epinephrine 1:200,000
  Arms: Bipivacaine 0.5% with epinephrine
Drug: Normal Saline — (placebo for bupivacaine)
  Other Names: 0.7%NS
  Arms: Normal Saline

SUMMARY:
Will patients that receive injections of Marcaine into the uterine nerve via the uterosacral ligaments experience less pain postoperatively, need less narcotic pain medication and return to activities of daily living sooner.

DETAILED DESCRIPTION:
Gynecologists use paracervical blocks in the office for decreasing pain during office based procedures. Paracervical blocks, in the office, work by injecting the cervix with local anesthetic, typically lidocaine, at the area of the uterosacral ligaments. The uterosacral ligaments contain the uterine nerve, which branches off of levels T12-L2. By injecting the uterine nerve with the local anesthetic patients are better able to tolerate the procedure and have decreased pain post procedure. In the office, paracervical blocks are performed vaginally with injections at the 3 o'clock and 9 o'clock position of the cervix. The use of paracervical blocks by Chudnoff et al reviewed the effectiveness of paracervical blocks in office based procedures, however no one has evaluated the effectiveness of injecting the uterosacral ligaments under direct visualization with the camera that is placed into the abdomen during a robotic assisted gynecologic procedure. We propose that by injecting the uterosacral ligaments and thus the uterine nerve during robotic assisted hysterectomies with Marcaine (Bupivacaine 0.5% with epinephrine 1:200,000) we can offer patients superior pain relief. The onset of action with Marcaine is rapid and anesthesia is long lasting. The duration of anesthesia is significantly longer with Marcaine than any other commonly used local anesthetic. It has also been noted that there is a period of analgesia that persists after the return of sensation, during which time the need for strong analgesics is reduced. By injecting Marcaine we hypothesize that patients will have decreased pain and need less narcotic pain medication. This will allow the patient to return to normal activities of daily living sooner.

This is a randomized controlled double blinded trial in which patients will be assigned to receive saline (control group) or bupivacaine 0.5% with epinephrine 1:200,000 (treatment group). The randomization will be performed through a computerized system in the pharmacy at the pharmacy of the hospital where the study is occurring. The randomization will occur once the patient has consented to the study. The treatment arm of the study will receive a total injection of 14ml of bupivacaine with 7ml directed into the right uterosacral ligament and 7ml into the left uterosacral ligament. The control arm of the study will receive a total injection of 14ml of normal saline with 7ml directed into the right uterosacral ligament and 7ml into the left uterosacral ligament. These injections will take place after the uterus and cervix have been surgically removed and the vaginal cuff has been surgically closed.

The maximum dose of bupivacaine with epinephrine is 225mg. The total amount of bupivacaine that we have chosen to inject is below the maximum allowable dosing and yet we believe will be an adequate amount for providing pain relief.

Eligible patients will be consented for the study while in the preoperative holding area. Once consented the patient will be given a medication diary form that they will take home. The form asks the patient to fill in the name of pain medication that they were prescribed and the dosage. They will also have an area for them to tally the number of pills they have taken since being discharged from the hospital. If they take anything for pain other than that prescribed by the physician who performed the surgery the patient will be taken out of the study. The Wong-baker faces pain rating scale is included on the form which they will be using to rate their pain during the telephone encounters.

The pharmacy will be notified once consent is obtained that the patient is participating in the study. After which, the injectable solution will be sent to the OR labeled "Study Drug." The surgical team and the patient will be blinded to which arm they are assigned to. With the use of a Bierman needle the solution will be injected into the uterine nerve as it courses with the uterosacral ligaments on each side at the level of the vaginal cuff. If the uterosacral ligaments cannot be easily identified, the patient will be excluded from the study.

Follow up will take place via telephone encounters.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotically assisted total hysterectomies with cystoscopy and with or without procedures involving the adnexa (salpingectomies and salpingo-oophorectomies)

Exclusion Criteria:

* Patients undergoing single incision procedures, those having supracervical hysterectomies and additional procedures involving their pelvic floor (including bladder neck suspension, anterior colophorraphy, posterior colophorraphy, perinealplasty) and sacracolpopexy
* Patients with allergies to bupivacaine and its derivatives
* Patients taking monoamine oxidase inhibitors or tricyclic antidepressants
* Patients with known clinically significant hepatic, gastrointestinal, renal, haematological, urologic, neurological, respiratory, endocrine or cardiovascular system abnormalities
* Patients with abnormal ECG's and prolonged QT syndrome
* Patients who are currently requiring narcotic pain medication or use narcotic pain medications regularly (more than twice weekly)

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pain scores using wong-baker faces pain rating scale | Post-operative day 1 or post-operative day 2 if they stay overnight following their surgery
  Follow up will take place via telephone encounters on post-operative day number one, unless the patient is admitted overnight following the surgery which in that case the telephone encounters will take place on postoperative day two. The patient will be asked to rate their average pain score for that day using the Wong-Baker faces pain rating scale which will occur at the time of the phone encounter.

SECONDARY OUTCOMES:
Type and amount of narcotic pain medication used to achieve pain relief | Post-operative day number one and five. Post-opertive day two and six if they stay overnight following their surgery
  The type and amount of narcotic pain medication used to achieve pain relief which will be documented using the medication diary given to patients prior to discharge home from the hospital.
Pain compared to a prior laparoscopic or robotic surgery | Post-operative day one and five, post-operative day two and six if they stay overnight in the hospital following their surgery
  Patient will be asked if they have ever had a laparoscopic or robotic surgery before and if they have how does their current pain with this surgery compare to their previous surgery. They will choose from the following answer choices: Worse, Better, No difference, Can not Recall.
Ability to drive | Post-operative day five, Postopertive day six if they stay overnight in the hospital following their surgery
  Patient will be asked if they have been able to drive since their surgery. If they have been able to drive we will ask how many days after surgery were they able to start driving.
Ability to perform household duties | Post-operative day five, Posoperative day six if they stay overnight in the hospital following their surgery
  On postoperative day five patient will be asked if they have been able to perform household duties. If their answer is yes they will then be asked how man days after their surgery were they able to start performing household duties
Ability to perform routine activities of daily living | Post-opertive day five, Postopertive day six if they stay overnight in the hospital following their surgery
  Patient will be asked if they have begun performing activities of daily living (i.e grooming, hygiene care, preparing meals). If patient says yes we will follow up asking the patient how many days after their surgery were they able to perform routine activities of daily living.
Body Mass Index | Obtained at time of admission to hospital
  Patient will be weighed upon admission to the hospital and asked what their height is at which time a BMI will be calculated.
Secondary pain scores using wong-baker faces pain rating scale | Post-operative day 5 or post-operative day 6 if they stay overnight following their surgery
  The second follow up will take place via telephone encounters on post-operative day number five, unless the patient is admitted overnight following the surgery which in that case the telephone encounters will take place on postoperative days six. The patient will be asked to rate their average pain score for that day using the Wong-Baker faces pain rating scale which will occur at the time of the phone encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Souza, DO, Principal Investigator — Souza, Amanda, M.D.
Locations (1):
- Botsford General Hospital, Farmington Hills, Michigan, United States

REFERENCES:
- [Background] Chudnoff S, Einstein M, Levie M. Paracervical block efficacy in office hysteroscopic sterilization: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):26-34. doi: 10.1097/AOG.0b013e3181c51ace. PMID 20027030